CLINICAL TRIAL: NCT06544564
Title: A Multi-Center, Prospective, Randomized Trial Evaluating the Efficacy of Membrane Wrap, A Human Amniotic Membrane on Venous Leg Ulcers in an Elderly Population
Brief Title: Human Amniotic Membrane On Venous Leg Ulcers In an Elderly Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioLab Holdings (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT-001-24
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 2 parallel groups randomly assigned in a 1:1 fashion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1- Membrane-Wrap™ plus SOC (Experimental): Membrane-Wrap ™ plus SOC Group 1 plus SOC treatment will be defined as: 1) debridement of non-viable, necrotic tissue, 2) application of Biologic as the primary, wound covering, 3) application of a dressing over Biologic that maintains moisture balance, 4) application of a Class 3 high compression system. A Class 3 high-compression system is required. High compression is useful for bigger legs or more active patients. High compression wraps can be used over padding on their own or as part of a layered system and should be applied in a spiral according to manufacturer's instructions. High strength compression can be applied successfully using many methods including but not limited to multilayered elastic compression, inelastic compression, Unna's boot, compression stockings, and other
  Interventions: Device: Membrane Wrap™
- Group 2: SOC only (Other): Group 2: Standard of Care only- Subjects randomized to Group 5 (SOC, or Active Control treatment) will not receive Biologic, but will receive SOC alone. SOC) is defined as: Compression treatment per Wound Healing Society guidelines, "Compression for treatment of Venous Ulcers" [10].
  SOC, or Active Control treatment, is defined as: 1) debridement of non-viable, necrotic tissue, 2) application of a primary, wound contact dressing that maintains moisture balance, 3) application of a Class 3 high compression system, and 4) wrapping with a covering, tertiary dressing. A Class 3 (most supportive) high-compression system is required. High compression bandages provide and maintain high levels of compression pressures in the range 25-35 mm Hg at the ankle. High strength compression can be applied successfully using many methods including multilayered elastic compression, inelastic compression, Unna's boot, compression stockings, and other.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Membrane Wrap™ — Membrane Wrap™
  Arms: Group 1- Membrane-Wrap™ plus SOC
Other: Standard of Care — SOC treatment will be defined as: 1) debridement of non-viable, necrotic tissue, 2) application of Biologic as the primary, wound covering, 3) application of a dressing over Biologic that maintains moisture balance, 4) application of a Class 3 high compression system, and 5) wrapping with a covering dressing
  Arms: Group 2: SOC only

SUMMARY:
This study is designed to assess the clinical effectiveness of Membrane Wrap, a human amniotic membrane for the management of difficult to heal partial- or full-thickness venous leg ulcers (VLUs)

DETAILED DESCRIPTION:
Multi-center (up to 20 sites), prospective, randomized trial assess the clinical effectiveness of human amniotic membrane(s) for the management of difficult to heal partial- or full-thickness venous leg ulcers (VLUs). The primary objective is to evaluate the effectiveness of Membrane wrap™ versus Standard of Care (SOC) in subject with eligible venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, subjects must meet all of the following criteria:

1. Ulcers of venous origin, as determined by clinical signs and symptoms (e.g. hyperpigmentation of the surrounding skin, history of swelling, varicosities, lipodermatosclerosis and/or dermatitis) or other assessments (e.g. venous reflux test). If the subject has multiple on the same leg and/or bilateral ulcers, the largest should be selected.
2. Venous insufficiency ulcers, of at least 1-month duration, which have not adequately responded to conventional ulcer therapy
3. Venous insufficiency ulcers between 2 cm2 and 16 cm2
4. Venous ulcer has not reduced in area ≥40% from baseline measurements during the 2-week screening period
5. Partial- or full-thickness VLU, including ulcers with tissue damage that extends through the epidermis and into the upper epidermis (papillary dermis), or into the deep dermis
6. Subjects are between 50 and 85 years of age.
7. Subject is expected to be available for 12-week follow-up
8. Subject, or their Legally Authorized Representative (LAR), has read, understood, and signed the IRB/IEC approved Informed Consent Form before screening procedures are undertaken.

Subjects who meet any of the following criteria will be excluded from participating in this study:

1. Ankle Brachial Index (ABI) of <0.7 or Toe Brachial Index (TBI) <0.5
2. Vasculitis, severe rheumatoid arthritis, and other collagen vascular diseases
3. Clinically significant medical conditions which would impair wound healing, as determined by the investigator, including renal, hepatic, hematologic, neurologic or immune disease
4. Signs and symptoms of infection, cellulitis, osteomyelitis
5. Necrotic ulcer beds
6. Subjects receiving hemodialysis or have uncontrolled diabetes: defined as A1C of greater than or equal to 12. An existing A1C value is allowed if completed within 3 months of subject screening.
7. Subjects who are currently receiving or have received at any time within one month prior to entry into the study, corticosteroids (>15 mg/day), immunosuppressive agents, radiation therapy, or chemotherapy. Anticipated use of the above agents will exclude subjects from entry into the study.
8. Wound unable to be debrided or subject not able to tolerate debridement
9. Subject not willing or able to comply with compression requirements
10. Subjects enrolled in other wound investigational studies within the past three months, or device studies within the past 30 days.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Time to wound closure by or on week 12. | 12 weeks
  Wound Closure is defined as:
  * Full epithelialization of the wound with the absence of drainage
  * Epithelialization is defined as a layer of epithelium visible on the wound surface
Frequency of wound closure by or on week 12. | 12 weeks
  Wound Closure is defined as:
  * Full epithelialization of the wound with the absence of drainage
  * Epithelialization is defined as a layer of epithelium visible on the wound surface

SECONDARY OUTCOMES:
Rate of VLU improvement by or on End of Study (EOS) from baseline | 12 weeks
  defined by:
  * >60% reduction in area, or
  * >60% reduction in depth, or
  * >75% reduction in volume Rate of VLU improvement by or on End of Study (EOS) from baseline

OTHER OUTCOMES:
Incidence of ulcer recurrence within the 12-week study period | 12 weeks
  Incidence of ulcer recurrence within the 12-week study period
Mean number of ulcer free days within the 12-week study period | 12 weeks
  Mean number of ulcer free days within the 12-week study period

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Medley, Study Chair — Sponsor GmbH
Locations (9):
- United States (9):
  - Tital Clinical Research, Mesa, Arizona
  - Center for Clinical Research, San Francisco, California
  - Midland Florida Clinical Research Center, DeLand, Florida
  - Biophase Research, North Miami Beach, Florida
  - Doctors Research Network, South Miami, Florida
  - Gateway Clinical Trials, O'Fallon, Illinois
  - Northwell Health, Lake Success, New York
  - Kent State College of Podiatry, Cleveland, Ohio
  - Advantage Foot Care of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No